### **Clinical Trial Protocol: CYS-004**

**Protocol Title:** A Phase 3, multi-center, randomized, double-masked,

vehicle-controlled clinical trial to assess the efficacy and safety of topical CyclASol® for the treatment of Dry Eye

Disease

**Protocol Number:** CYS-004 / ESSENCE 2

Trial Phase: 3

**Investigational Product Name:** CyclASol® 0.1 % Ophthalmic Solution (Cyclosporine A

0.1%)

**IND Number:** 128163

**Indication:** Dry Eye Disease (*keratoconjunctivitis sicca*)

**Sponsor:** Novaliq GmbH

Im Neuenheimer Feld 515

69120 Heidelberg

Germany

**Contract Research Organization:** 



Original Protocol: 27<sup>th</sup> August 2020 Amendment 1: 2<sup>nd</sup> December 2020 Amendment 2: 15<sup>th</sup> March 2021

### **Confidentiality Statement**

This protocol contains confidential, proprietary information of and Novaliq GmbH. Further dissemination, distribution, or copying of this protocol or its contents is strictly prohibited.

### **Regulatory Statement**

This trial will be performed in compliance with the protocol and in accordance with Good Clinical Practice (International Conference on Harmonisation [ICH], Guidance E6), principles of human subject protection, and applicable country-specific regulatory requirements.


### 1 SYNOPSIS AND TRIAL CONTACT INFORMATION

### 1.1 TRIAL CONTACT INFORMATION

### **SPONSOR PERSONNEL**

| Scientific Lead: | _ |
|----------------------|---|
| Clinical Operations: | |

### **MEDICAL MONITOR**

| | _ |
|-----------------|---|
| Medical Monitor | |

## PERSONNEL

| Clinical Project Manager: | - |
|---------------------------|---|
| Biostatistician: | |


### 1.2 SYNOPSIS

| Protocol Title: | A Phase 3, multi-center, randomized, double-masked, vehicle-controlled clinical trial to assess the efficacy and safety of topical |
|---|---|
| | CyclASol® for the treatment of Dry Eye Disease |
| Protocol Number: | CYS-004 / ESSENCE 2 |
| Investigational Medicinal Product: | <ol> <li>CyclASol 0.1% Ophthalmic Solution (Cyclosporine A 0.1% solution)</li> <li>Vehicle Ophthalmic Solution (F4H5)</li> </ol> |
| Trial Phase: | 3 |
| That Fliase. | The objective of this trial is to assess the efficacy, safety, and |
| Trial Objective | tolerability of CyclASol 0.1% Ophthalmic Solution in comparison to the vehicle for the treatment of the signs and symptoms of Dry Eye Disease (DED). |
| Overall Trial Design: | |
| Structure: | This clinical trial is multi-center, randomized, double-masked, and vehicle-controlled with a run-in period with artificial tears. |
| Participant Duration: | An individual subject's participation is estimated to be approximately 6 weeks (approx. 2 weeks screening and 4 weeks treatment period). |
| Trial Duration | The estimated trial duration is 8 months, from first subject first visit to last subject last visit. |
| Controls: | Vehicle (F4H5) |
| Dosage/Dose Regimen: | <ul> <li>Eligible subjects will be randomized to one of the following treatments to be administered BID bilaterally for approximately 29 days (from Visit 1 to Visit 3).</li> <li>CyclASol 0.1% Ophthalmic Solution (Cyclosporine A 0.1% solution)</li> <li>Vehicle (F4H5)</li> <li>A 14-day run-in period will be used for subject selection before randomization. During this period, all subjects will receive Systane® Balance to administer bilaterally BID.</li> </ul> |
| Summary of Visit<br>Schedule: | <ul> <li>4 visits over the course of approximately 6 weeks:</li> <li>Visit 0, Day -14 ± 2 days, Screening;</li> <li>Visit 1, Day 1, Baseline/Randomization;</li> <li>Visit 2, Day 15 ± 2 days, 2-Week Follow-Up;</li> <li>Visit 3, Day 29 ± 2 days, 4-Week Follow-Up and Trial Exit</li> </ul> |
| Measures Taken to | This is a multi-center, randomized, double-masked and vehicle- |
| Reduce Bias: | controlled clinical trial. |
| Trial Population Characte | ristics: |
| Number of Subjects: | Approximately subjects will be screened to enroll at least 834 (417 per treatment arm) subjects at approximately 25 sites. |
| Condition/Disease: | Dry Eye Disease (keratoconjunctivitis sicca) |
| Inclusion Criteria: | Each subject must: |
| | 1. Be at least 18 years of age; |


| | 2. | Provide written informed consent; |
|---|---|---|
| | 3. | Have a subject reported history of Dry Eye Disease |
| | 4. | Be currently using or have used over-the-counter (OTC) |
| | | eye drops, lubricating gels, nerve stimulation devices for |
| | | tear productions (e.g. TrueTear <sup>TM</sup> ) and/or artificial tears |
| | | for dry eye symptoms within 30 days before Visit 0; |
| | 5. | Have a Dryness Score |
| | | Have a total corneal fluorescein staining (tCFS) score of |
| | | Time we were the second state of the second st |
| | 7 | Have a total lissamine green conjunctival score |
| | , · | Thave a total hosailine green conjunctival score |
| | 8 | Have an unanesthetized Schirmer's Test score |
| | 0. | Thave an analicstrictized Schiffier 5 Test score |
| | 9. | |
| | J. | |
| | 10 | . Be able and willing to follow instructions and participate |
| | 10 | in all trial assessments and visits. |
| <b>Exclusion Criteria:</b> | Each | subject must not: |
| L'Actusion Cificilia. | | Have any clinically significant slit-lamp findings at Visit |
| | 1. | Thave any entire any significant site famp intenings at visit |
| | | 0 that require prescriptive medical treatment and/or in the |
| | | 0 that require prescriptive medical treatment and/or in the opinion of the investigator may interfere with trial |
| | | opinion of the investigator may interfere with trial |
| | | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, |
| | 2 | opinion of the investigator may interfere with trial |
| | 2. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, |
| | | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, |
| | 2. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, |
| | 3. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, advanced epithelial basement membrane disease; |
| | 3. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, advanced epithelial basement membrane disease; Have abnormal lid anatomy (e.g. incomplete eyelid |
| | 3.<br>4. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, advanced epithelial basement membrane disease; |
| | 3. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, advanced epithelial basement membrane disease; Have abnormal lid anatomy (e.g. incomplete eyelid |
| | 3.<br>4. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, advanced epithelial basement membrane disease; Have abnormal lid anatomy (e.g. incomplete eyelid |
| | 3.<br>4. | opinion of the investigator may interfere with trial parameters including trauma, Stevens-Johnson Syndrome, advanced epithelial basement membrane disease; Have abnormal lid anatomy (e.g. incomplete eyelid |


| <br> |
|---------------------------------------------------------------|
| 7. |
| 8. Have a history of herpetic keratitis; |
| 9. Have active ocular allergies or ocular allergies that may |
| become active during the trial period; |
| 10. Have worn contact lenses within 90 days before Visit 0 or |
| anticipate using contact lenses during the trial; |
| 11. |
| 12. Be diagnosed with an ongoing ocular infection; |
| 22. Have an ongoing systemic infection (bacterial, viral, or |
| fungal), including a fever, and/or requiring treatment with |
| antibiotics at Visit 0 or Visit 1 and/or positive SARS-CoV- |
| 2 (COVID-19) test within 2 weeks before Visit 0 and until |
| Visit 1; |


### **Key Secondary Efficacy Endpoints:**

- CFB in total conjunctival lissamine green staining score (Oxford scale) at Day 29
- Proportion of responders in central corneal fluorescein staining (cCFS) score (≥ 1 score improvement on NEI scale) at Day 29
- Proportion of responders in tCFS score (≥ 3 score improvement on NEI scale) at Day 29
- CFB in cCFS score (NEI scale) at Day 29
- CFB in tCFS (NEI scale) at Day 15
- CFB in visual analogue scale (VAS) for blurred vision at Day
   29




# Visual acuity and CFB at each measured post-baseline visits; Slit-lamp biomicroscopy findings and CFB at each measured post-baseline visits Intraocular pressure and CFB at each measured post-baseline visits Dilated fundoscopy findings and CFB at each measured post-baseline visits Systemic and ocular AEs

### **General Statistical Methods and Types of Analyses**

### Sample Size:

The trial has been designed to have 90% power assuming independence between the sign and symptom primary efficacy endpoints; positive correlation between these two endpoints would increase the overall power. Accounting for subject discontinuations, approximately 834 total subjects (417 per treatment arm) will be enrolled assuming a dropout rate of approximately 10%.

### **Multiplicity Considerations:**

Hierarchical fixed sequence testing will be employed to maintain the type I error rate. The primary analyses will first test the difference in the mean CFB corneal fluorescein staining (NEI scale) total score between treatments at Day 29. If the test of the difference is statistically significant at the two-sided alpha = 0.05 level in favor of CyclASol, then the trial will be considered a success; CyclASol will be declared to be superior to vehicle in the mean CFB corneal fluorescein staining (NEI scale) total score at Day 29; and the difference in the mean CFB Dryness Score (VAS) between treatments at Day 29 will be tested at the two-sided alpha = 0.05 level.

If in addition to a statistically significant test of the difference in the mean CFB tCFS score (NEI scale) at Day 29 in favor of CyclASol, the test of the difference in the mean CFB Dryness Score (VAS) at Day 29 is also statistically significant in favor of CyclASol, then CyclASol will be declared to be superior to vehicle in both the mean CFB tCFS score (NEI scale) and the mean CFB Dryness Score (VAS) at Day 29.

### Primary Efficacy Analyses:

The primary comparisons in this trial will be between CyclASol versus vehicle at Day 29. The primary efficacy endpoint (e.g. CFB in tCFS) will be summarized descriptively (n, mean, standard deviation, median, min, and max) and analyzed using an ANCOVA model with terms for baseline value and treatment.

Least squares mean for each treatment group and for the difference between treatment groups will be presented from the model together with two-sided p-values and 95% confidence intervals.

The primary analysis will use the Full Analysis Set (FAS) with available data per subject using Estimand 1, assuming the rate of missing data for an endpoint is <5%. If the rate of missing data for an endpoint is  $\ge5\%$  and the missing data is:

1. Balanced between treatment groups, then the primary analysis will be based on the primary multiple imputation methodology as presented in Estimand 2 and the available data analyses will become robustness analyses.


2. Imbalanced between treatment groups, then the primary analysis will be based on trimmed means (Permutt et al., 2017) as presented in Estimand 3 and the available data analyses will become robustness analyses.

Two-sample t-tests, Wilcoxon rank sum tests and mixed-effect repeated measures analysis comparing treatment groups will be performed as sensitivity analyses.

Additional sensitivity analyses will include repeating the primary analysis on the FAS imputing missing data using multiple imputation methodology under different assumptions of missingness (at random and not at random); last observation carried forward (LOCF); trimmed means as specified in Estimand 3; and the per protocol set (PPS) with available data per subject. Sensitivity analyses will also include repeating the primary analysis using the FAS with multiple imputation methology and different assumptions for intercurrent events due to COVID-19.

### Secondary Efficacy Analysis:

The following key secondary endpoints will be tested hierarchically:

- 1. CFB in total conjunctival lissamine green staining score (Oxford scale) at Day 29
- 2. Proportion of responders in cCFS score (≥ 1 score improvement on NEI scale) at Day 29
- 3. Proportion of responders in tCFS (≥ 3 score improvement on NEI scale) at Day 29
- 4. CFB in cCFS score (NEI scale) at Day 29

Inference will only be made on these endpoints, at a 2-sided alpha = 0.05, if both primary endpoints and any higher order key secondary endpoints are statistically significant at a 2-sided alpha = 0.05 in favor of CyclASol.

If all four of these key secondary endpoints and both primary endpoints demonstrate statistical significance at a 2-sided apha = 0.05 in favor of CyclASol, then the following two key secondary endpoints will be tested simultanteously using Hochberg's procedure to maintain an overall two-sided alpha = 0.05:

- CFB in visual analogue scale (VAS) for blurred vision and at Day 29
- CFB in tCFS (NEI scale) at Day 15

Quantitative key secondary efficacy endpoints will be analyzed (similar ANCOVA model) and summarized similarly to the primary effiacy endpoints. Dichotomous key secondary endpoints (proportion of responders) will be summarized descriptively (frequency and percentage) and analyzed using a logistic regression model with terms for baseline value and treatment.

### Safety Variables

Adverse events (AEs) will be coded using the MedDRA dictionary. Frequencies and percentages of treatment-emergent adverse events (TEAEs) will be summarized at the subject level by system organ class and preferred term for all TEAEs, treatment related TEAEs, serious TEAEs, and TEAEs causing premature discontinuation by treatment group. Other safety endpoints including visual acuity, slit-lamp biomicroscopy findings, intraocular pressure, and dilated fundoscopy will be summarized by treatment group and visit using descriptive statistics.


# TABLE OF CONTENTS SYNOBSIS AND TRIAL

| 1 | SYN | OPSIS AND TRIAL CONTACT INFORMATION2 |
|---|---|---|
| | 1.1 | TRIAL CONTACT INFORMATION 2 |
| | 1.2 | SYNOPSIS |
| | | OF CONTENTS10 |
| | | ABBREVIATIONS |
| 2 | INTI<br>2.1 | RODUCTION 15 Dry Eye Disease (DED) 15 |
| | 2.1 | Product Rational |
| | 2.3 | Trial Rational |
| | 2.4 | Summary of Known and Potential Risks and Benefits to Human Subjects 16 |
| 3 | | AL OBJECTIVES |
| | 3.1 | Primary objective |
| | 3.2 | Secondary objectives |
| 4 | TRIA<br>4.1 | AL DESIGN |
| | | Overall Trial Design |
| | 4.2 | End of Trial Definition |
| | 4.3 | Visit Description |
| | 4.4 | Trial Flow |
| | 4.5 | Enrollment and Treatment Assignment |
| | 4.6 | Justification of Trial Design20 |
| | 4.7 | Justification for Dose |
| 5 | | AL POPULATION21 |
| | 5.1 | Number of Subjects (approximate)21 |
| | 5.2 | Trial Population Characteristics21 |
| | 5.3 | Inclusion Criteria |
| | <b>5.4</b> | Exclusion Criteria |
| | 5.5 | Subject/ Trial Withdrawal Criteria24 |
| 6 | TRIA | AL PARAMETERS25 |
| | 6.1 | Efficacy Endpoints |
| | | 6.1.1 Primary Efficacy Endpoints |
| | | 6.1.2 Key Secondary Efficacy Endpoints |
| | 6.2 | Safety Endpoints |
| | 6.3 | |
| 7 | | AL MATERIALS27 |
| ′ | 7.1 | Investigational Medicinal Product(s) |
| | | 7.1.1 IMP(s)/ Formulation(s) |

| | | 7.1.2 Labeling and Packaging of IMP | 27 |
|---|---|---|---|
| | | 7.1.3 IMP Storage | 28 |
| | | 7.1.4 Administration of run-in medication | |
| | | 7.1.5 IMP Dispensation | |
| | <i>7</i> 2 | 7.1.6 Instructions for Use and Administration | |
| | 7.2 | IMP Accountability | |
| | 7.3 | IMP Handling and Disposal | |
| | 7.4 | Other Trial Supplies | |
| 8 | | AL METHODS AND PROCEDURES | |
| | 8.1 | Concurrent Medications and Therapies | |
| | 8.2 | Prohibited Medications | 30 |
| | 8.3 | Restrictions and Prohibitions | 30 |
| | 8.4 | Examination Procedures | 31 |
| | | 8.4.1 Procedures to be performed at Each Trial Visit with Regard to Trial Objective(s) | 31 |
| | | 8.4.2 Early Termination/Discontinuations | |
| | | 8.4.3 Unscheduled Visits | |
| | 8.5 | Compliance with Dosing/Protocol Deviations | 34 |
| | 8.6 | Subject Disposition | 35 |
| | | 8.6.1 Completed Subjects | 35 |
| | | 8.6.2 Discontinued Subjects | |
| | <b>8.7</b> | Trial Termination | 35 |
| | 8.8 | Trial Duration | 36 |
| 9 | ADV | ERSE EVENTS | 37 |
| | 9.1 | Adverse Event | 37 |
| | | 9.1.1 Severity | 37 |
| | | 9.1.2 Relationship to Investigational Product | |
| | | 9.1.3 Expectedness | |
| | | 9.1.4 Outcome | |
| | 9.2 | 9.1.5 Period of Observation | |
| | 9.3 | Procedures for Reporting Adverse Events | |
| | 9.3 | • | |
| | | <ul><li>9.3.1 Reporting a Serious Adverse Event</li><li>9.3.2 Reporting a Suspected Unexpected Serious Adverse Reaction</li></ul> | |
| | 9.4 | Procedures for Unmasking of IMP | |
| | 9.5 | Type and Duration of the Follow-up of Subjects after Adverse Events | |
| | 9.6 | Procedures for Reporting Pregnancies | |
| 10 | | | |
| 10 | 10.1 | TISTICAL HYPOTHESES AND METHODS OF ANALYSESAnalysis Populations | |
| | | • • | |
| | 10.2 | Statistical Hypotheses | |
| | 10.3 | Sample Size | 44 |

| | 10.4 | Statistical Analysis | 44 |
|---|---|---|---|
| | | 10.4.1 General Considerations | 44 |
| | | 10.4.2 Unit of Analysis | 45 |
| | | 10.4.3 Missing Data | 45 |
| | | 10.4.4 Multiplicity Considerations | |
| | | 10.4.5 Primary Efficacy Analyses | |
| | | 10.4.6 Key Secondary Efficacy Analyses | 50 |
| | | 10.4.7 | |
| | | 10.4.8 | 5.1 |
| | | 10.4.9 Safety Variables Analyses | |
| | 10.5 | Additional Analyses | |
| 11 | | IPLIANCE WITH GOOD CLINICAL PRACTICES, ETHICAL | |
| COI | | CRATIONS, AND ADMINISTRATIVE ISSUES | 53 |
| | 11.1 | Protection of Human Subjects | 53 |
| | | 11.1.1 Subject Informed Consent | 53 |
| | | 11.1.2 Institutional Review Board (IRB) Approval | |
| | 11.2 | Ethical Conduct of the Trial | 53 |
| | 11.3 | Subject Confidentiality | 54 |
| | 11.4 | Documentation | 54 |
| | | 11.4.1 Retention of Documentation | 54 |
| | 11.5 | Recording of Data on Source Documents and Electronic Case Rep | orts Forms |
| | | (eCRFs) | 55 |
| | 11.6 | Monitoring and Quality Assurance | 55 |
| | 11.7 | Handling of Biological Samples | 55 |
| | 11.8 | Publications | 55 |
| 12 | REF | ERENCES | 56 |
| App | | 1: Schedule of Assessments | |
| App | endix | 2: Examination Procedures, Tests, Equipment, and Techniques | 59 |
| App | endix | 3: Protocol Amendment Summary | 75 |
| | Ame | ndment 1 | 75 |
| | Ame | ndment 2 | 77 |
| App | endix | 4: Change History | 85 |
| | | 5: Sponsor and CRO Approvals | |
| App | endix | 6: Investigator's Signature | 87 |

### LIST OF ABBREVIATIONS

AE Adverse Event

AlCc Akaike Information Criterion with a correction for finite

sample sizes

ANCOVA Analysis of Covariance
BCVA Best-Corrected Visual Acuity

BID Twice Daily

BLQ Below the Limit of Quantification cCFS Central corneal fluorescein staining

CFB Change from Baseline
CFR Code of Federal Regulations
CFS Corneal fluorescein staining

CI Confidence Interval

CRA Clinical Research Associate
eCRF Electronic Case Report Form
CRO Contract Research Organization

CS Compound Symmetry

CsA Cyclosporine A
CV Curriculum Vitae
DED Dry Eye Disease

DEWS (International) Dry Eye Workshop

ECG Electrocardiography, Electrocardiogram

ET Early Termination

ETDRS Early Treatment of Diabetic Retinopathy Study

FAS Full Analysis Set

FDA Food and Drug Administration

g Gram

GCP Good Clinical Practice
GMP Good Manufacturing Practice

HIPAA Health Information Portability and Accountability Act

IB Investigators' Brochure

ICH International Conference on Harmonization

IEC Independent Ethics CommitteeIMP Investigational Medicinal ProductIND Investigational New Drug Application

IOP Intraocular Pressure

IRB Independent Review Board

IRT Interactive Response Technology

IUD Intrauterine Device

LOCF Last Observation Carried Forward

logMAR Logarithm of the Minimum Angle of Resolution

MCMC Markov Chain Monte Carlo

MedDRA Medical Dictionary for Regulatory Activities


MGD Meibomian Gland Dysfunction

 $\begin{array}{ccc} mL & & Milliliter \\ \mu L & & Microliter \\ mm & & Millimeter \end{array}$ 

mmHg Millimeters of Mercury

NCS Not Clinically Significant
NDA New Drug Application
NEI National Eye Institute

NONMEM Non-linear mixed effects modeling

OD Right Eye
OS Left Eye

OSDI Ocular Surface Disease Index

OU Both Eyes

OTC Over the Counter PPS Per Protocol Set

SAE Serious Adverse Event

SAF Safety Set

SFA Semifluorinated Alkane

SOP Standard Operating Procedures tCFS Total corneal fluorescein staining TEAE Treatment-emergent Adverse Event

TFBUT Tear Film Break-up Time

TMF Trial Master File

US(A) United States (of America)

VA Visual Acuity

VAS Visual Analog Scale

WHO World Health Organization

w/v Weight per volume w/w Weight per weight


### 2 INTRODUCTION

### 2.1 Dry Eye Disease (DED)

Dry Eye Disease (DED) is defined by the International Dry Eye Workshop (DEWS) as a multifactorial disease of the ocular surface characterized by a loss of homeostasis of the tear film, and accompanied by ocular symptoms, in which tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neurosensory abnormalities play etiological roles (Craig et al. 2017). Symptoms of DED such as feeling of dryness, burning, a sandy/gritty sensation, foreign body sensation, pain or itchiness are quite debilitating. In addition, visual function related symptoms such as fluctuating vision with blinking, blurred vision, and difficulty with reading despite perfect visual acuity is an important and underestimated aspect of the disease. In consequence, DED negatively impacts quality of life comparably to other severe diseases (Schiffman et al. 2003), and adverse effects on mental health, such as depression and anxiety, have been observed (Le et al. 2012). DED is a serious disorder that, if left untreated or undertreated, progressively damages the ocular surface and may lead to vision loss due to corneal complications (Lemp et al. 1995).

As many as 5 - 35% of subjects visiting ophthalmic clinics report dry eye symptoms, making it one of the most common conditions seen by ophthalmic specialists (McCarty et al. 1998; Lin et al. 2003). Estimates of the prevalence of dry eye vary considerably, depending on the criteria used to define the disease, but in the United States (US), it has been estimated that as many as 3.2 million women and 1.7 million men over the age of 50 have DED, with a projected 40% increase in the number of patients affected by 2030 (Schaumberg et al. 2002; Schaumberg et al. 2003; Schaumberg et al. 2009) With the aging population in the US and other countries of the developed world, and with increasing use of visual displays / computers, DED is expected to continue to become more prevalent and finding a treatment is becoming more important (Benitez-del-Castillo et al. 2017).

### 2.2 Product Rational

Cyclosporine A (CsA), a potent and selective immunomodulatory drug, acts as a regulator of T-cells via inhibition of calcineurin. Due to this mode of action it has been widely studied as topical treatment for T-cell mediated diseases of the ocular surface such as DED. In the US, CsA eye drops formulated as an emulsion have been approved and marketed as Restasis 0.05% for this indication since 2002. In Europe, Ikervis<sup>TM</sup>, a 0.1% CsA emulsion formulation, received a marketing authorization by the European Medicines Agency for the treatment of DED in early 2015. A second CsA containing product, Cequa<sup>TM</sup>, a nano-emulsion was approved in the US in 2018.

CyclASol, in contrast, is a clear ophthalmic solution of CsA developed with the goal of avoiding the use of oils, surfactants and preservatives. Potential benefits from the CyclASol formulation include improved tolerability and efficacy, early onset of efficacy and decreased visual disturbances associated with oily eye drops, emulsions or ointments. Moreover, the multiple dose containers allow for a convenient handling.


solubilization of CsA in CyclASol, the semifluorinated alkane the F4H5is used as the vehicle. F4H5 is colourless, has a high vapor pressure, and is immiscible with water while having nearly the same refractory index. F4H5's physical properties make it an optimal vehicle for topical ocular use. As a result of its high vapor pressure (Krafft et al. 2009), F4H5 dissipates quickly from the ocular surface and consequently does not interact physically with the tear film, as shown in rabbits, where F4H5 had no effect on tear film break-up time (TFBUT) (Agarwal et al. 2019). Due to the low surface tension of F4H5, CyclASol eye drops are of small size, potentially reducing pre-corneal clearance. Importantly, the low surface tension of the CyclASol formulation facilitates dissemination of the applied eye drop on the conjunctiva. The dissemination and spreading properties are further thought to improve the local bioavailability.

### 2.3 Trial Rational

After successful preclinical testing and early clinical testing, a Phase 2b/3 clinical trial (CYS-003, ESSENCE) was recently completed confirming the effects seen in the Phase 2 clinical trial.

In CYS-003, CyclASol 0.1% met the primary sign endpoint, showing superiority compared to vehicle in change from baseline (CFB) in total corneal fluorescein staining (tCFS) at Day 29 with high statistical significance (p=0.0002). CyclASol 0.1% also showed trends of more improvement in the second primary endpoint of CFB in total OSDI<sup>©</sup> at Day 29. Additionally, a statistically significant greater improvement in the pre-specified secondary symptom endpoint CFB in "Dryness Score" (visual analogue scale for severity of dryness) at Day 29 was demonstrated in the CyclASol 0.1% treatment group compared to the vehicle group (p=0.0311).

Furthermore, the CyclASol 0.1% group consistently showed statistically significant improvements over time in corneal and conjunctival staining compared to vehicle. The clinical effects observed had an early onset after 14 days of treatment that continued over the 84-day treatment period.

This second pivotal Phase 3 trial is designed to replicate efficacy of CyclASol 0.1% BID dosing over vehicle as already demonstrated in CYS-003 (ESSENCE) on sign (CFB in tCFS) and symptom (CFB in Dryness Score) at Day 29. The trial will be powered to demonstrate efficacy of CyclASol 0.1% over vehicle in both endpoints. The trial will further investigate the safety and tolerability of CyclASol 0.1%.

### 2.4 Summary of Known and Potential Risks and Benefits to Human Subjects

The investigational medicinal product (IMP) CyclASol 0.1% Ophthalmic Solution contains CsA as active ingredient and its vehicle, which consists of F4H5. CsA is a potent and selective immunosuppressive drug, used routinely for decades as an oral immunomodulator in various indications. CsA containing eye drops have been proven safe over the last 15 years. The excipient F4H5 used in CyclASol is chemically inert, without pharmacologic activity and not undergoing metabolism in the human body. However, it is not part of any pharmaceutical product approved


so far. Therefore, it has been subjected to the same pivotal non-clinical studies as a new active substance with favorable results.

282 subjects have been exposed to CyclASol 0.05% or 0.1% for up to 4 months duration in clinical trials to date (clinical trials CYS-001: Phase 1; CYS-002: Phase 2; CYS-003: Phase 2b/3) with a favorable outcome in safety and tolerability.



In summary, based on the preclinical and clinical data obtained to date, risks to subjects in the planned CYS-004 trial are considered very low. Furthermore, the subjects randomized in the trial will be closely monitored, and current standard ophthalmic safety assessments will be performed during the entire treatment period. The results demonstrated to date the efficacy of CyclASol on signs and symptoms of DED. Treatment with CyclASol therefore provides a favorable benefit-risk


profile in subjects with DED, addressing a clinical need that is currently not optimally addressed with available treatment options for DED.

This clinical trial CYS-004 is designed to confirm the positive benefit-risk profile.

### 3 TRIAL OBJECTIVES

### 3.1 Primary objective

• The primary objective of the study is to assess efficacy of CyclASol in comparison to the vehicle for the treatment of a sign and symptom of DED.

### 3.2 Secondary objectives

• The secondary objective is to assess safety and tolerability of CyclASol in comparison to the vehicle for the treatment of signs and symptoms of DED.

### 4 TRIAL DESIGN

### 4.1 Overall Trial Design

This is a Phase 3 multicenter, randomized, double-masked, and vehicle-controlled clinical trial to evaluate the efficacy, safety and tolerability of CyclASol 0.1% Ophthalmic Solution in subjects with signs and symptoms of DED. Approximately 834 subjects of either sex and of any race who are at least 18 years of age with a subject-reported history of dry eye in both eyes and meeting all other trial eligibility criteria will be randomized at approximately 25 sites in the US to receive treatment with CyclASol or vehicle in a 1:1 ratio (approx. 417 subjects per treatment arm).

This trial is composed of two distinct parts: a run-in period and a treatment period. During the 14-day run-in period, subjects will dose Systane Balance bilaterally BID. Eligible subjects will thereafter dose the IMP (CyclASol or vehicle) bilaterally BID for approximately 29 days.

### 4.2 End of Trial Definition

The end of the trial for an individual subject is defined as that subject's last visit as specified in the Schedule of Assessments.

The end of the trial for the overall trial is defined as completion of the last visit or procedure as specified in Schedule of Assessments for all subjects in the trial.


### 4.3 Visit Description

Subjects will be required to sign an Informed Consent before completing any trial related procedure. All examination procedures are listed in Section 8.4 and in the Schedule of Assessments. For consistency and to avoid interference, they should be performed in the respective order as listed. Trial Drug Dispensation is described in Section 7.1.5.

### Screening (Visit 0)



### **Baseline** (Visit 1)



### Visits 2-3



### **Early Termination (ET)**

Subjects who terminate early during the treatment period will be asked to complete all assessments as indicated at Visit 3 on the schedule of assessments prior to commencement of any alternative dry eye therapy (if considered possible). Dosing diary and trial medication will be collected. Subjects who are terminated early from the trial will not be replaced.


### 4.4 Trial Flow



### 4.5 Enrollment and Treatment Assignment

All treatment arms will be enrolled in parallel. Each subject will be assigned a unique subject number. All subject numbers will be assigned in sequential order by the site using a two (2) digit site number and three (3) digit subject number format (XX-XXX). If all inclusion and none of the exclusion criteria are met at Visits 0 and 1, each qualifying subject will then be randomized.

The IRT will be used to account for the stratification factor while assigning the drug kit numbers at Visit 1. The

be used to account for the stratification factor while assigning the drug kit numbers at Visit 1. The subjects, investigators, personnel involved in conduct and monitoring of the trial and sponsor will be masked to IMP assignment.

Each subject will spend approximately 6 weeks in the trial. The total duration of the trial from "first subject in" to "last subject out" is expected to be approximately 8 months.

### 4.6 Justification of Trial Design

This trial is designed as a confirmatory trial to the previously conducted Phase 2b/3 trial CYS-003 in subjects with DED.

The trial will be a randomized, double-masked, vehicle-controlled trial to demonstrate efficacy and safety of CyclASol after 1-month treatment duration. Vehicle controlled clinical trials are currently the standard for DED trials. Randomization and double masking are state of the art measures to reduce bias. Fast onset of efficacy is important for subjects and their compliance to therapies, thus early demonstration of efficacy (e.g. at 1 month) is desired and highly clinically relevant. Moreover, DED is a fluctuating condition with phase-like recurring dry eye complaints that may be linked to seasonal and / or environmental changes (van Setten et al. 2016), thus a primary endpoint assessment at a shorter treatment duration is considered clinically relevant and has a greater potential to capture the true drug effect.

Total corneal fluorescein staining (NEI grading) and Dryness Score (VAS) have been selected as the primary sign endpoint and primary symptom endpoint, respectively. Corneal staining is an accepted clinical endpoint in DED and a highly relevant marker in this disease, as stained areas represent punctate disruption and damage of the corneal epithelium (Pflugfelder et al. 2017).


Reduction of corneal staining reflects corneal surface healing and thus is highly representative of treatment success. In DED trials, common symptoms such as dryness, frequency of dryness, blurred vision are frequently graded using the VAS (<u>Novack et al. 2017</u>). Questionnaires using VAS to assess symptoms of DED are generally considered validated symptom questionnaires in DED.

The two primary endpoints, CFB in tCFS and CFB in Dryness Score, will be tested in a hierarchical order with tCFS being tested first. The hierarchical testing has been selected to protect the  $\alpha$  – error.

### 4.7 Justification for Dose

The CyclASol 0.1% BID was selected for the first pivotal trial CYS-003 based on results of CYS-002. The aim of the current trial CYS-004 is to replicate the efficacy and safety results of CYS-003, consequently the same dose and dosing schedule will be tested.

### 5 TRIAL POPULATION

### 5.1 Number of Subjects (approximate)

An estimated subjects will be screened to randomly assign at least 834 subjects to IMP such that at least 379 evaluable subjects per treatment arm complete the trial.

### 5.2 Trial Population Characteristics

All subjects must be at least 18 years of age, of either sex, and of any race. Furthermore, subjects must have a subject-reported history of dry eye in both eyes and meet all inclusion criteria and none of the exclusion criteria.

### 5.3 Inclusion Criteria

Subjects will be eligible to participate in this trial if they **meet all** following criteria:

- 1. Be at least 18 years of age;
- 2. Provide written informed consent;
- 3. <u>Have a subject reported history of Dry Eye Disease</u>
- 4. Be currently using or have used over-the-counter (OTC) eye drops, lubricating gels, nerve stimulation devices for tear productions (e.g. TrueTear) and/or artificial tears for dry eye symptoms within 30 days before Visit 0;
- 5. Have a Dryness Score




8. Have a history of herpetic keratitis;

7.

9. Have active ocular allergies or ocular allergies that may become active during the trial period;


10. Have worn contact lenses within 90 days before Visit 0 or anticipate using contact lenses during the trial;

| 11. |
|-----|

- 12. Be diagnosed with an ongoing ocular infection;
- 13. Have had intraocular surgery or ocular laser surgery within 180 days before Visit 0, or have any planned ocular or eyelid surgeries during the trial period;
- 14. Have active ocular or periocular rosacea or a pterygium;



- 22. Have an ongoing systemic infection (bacterial, viral, or fungal), including a fever, and/or requiring treatment with antibiotics at Visit 0 or Visit 1 and/or positive SARS-CoV-2 (COVID-19) test within 2 weeks before Visit 0 and until Visit 1;
- 23. Have been randomized in a previous CyclASol trial;
- 24. Be a woman who is pregnant, nursing, or planning a pregnancy;
- 25. Be unwilling to submit a urine pregnancy test at Visit 0 and Visit 3 (or early termination visit) if of childbearing potential. Non-childbearing potential is defined as a woman who is permanently sterilized (i.e. has had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or is post-menopausal (i.e. without menses for 12 consecutive months);


- 26. Be a woman of childbearing potential who is not using an acceptable means of contraception. Acceptable methods of contraception include hormonal contraceptives (i.e. oral, implantable, injectable, or transdermal contraceptives), mechanical contraceptives (i.e. spermicide in conjunction with a barrier such as a diaphragm or a condom), intrauterine devices (IUD), or the surgical sterilization of the partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the trial, she must agree to use adequate birth control as defined above for the remainder of the trial;
- 27. Have an uncontrolled systemic disease;



30. Have a condition or be in a situation (e.g. language barrier, illiteracy) which the investigator feels may put the subject at significant risk, may confound the trial results, or may interfere with the subject's participation in the trial significantly.

### 5.5 Subject/ Trial Withdrawal Criteria

Subjects are free to discontinue their participation in the trial at any time without giving their reasons.

A subject **must be** discontinued after randomization **from the trial** for any of the following reasons:

- Occurrence of pregnancy;
- Withdrawal of subject's consent;
- Emergency unblinding has occurred.

A subject **must be** discontinued **from treatment** after randomization for any of the following reasons (but may remain in the trial for follow up assessments):

- If at any time during the trial the investigator determines that a subject's safety has been compromised;
- Occurrence of an exclusion criterion that is clinically relevant and affects the subject's safety as judged by the investigator and/or sponsor;
- If discontinuation is considered necessary by the investigator and/or sponsor;
- Occurrence of AEs that present an unacceptable consequence or risk to the subject in the judgment of the investigator, sponsor, or the medical monitor;


• If a subject has failed to attend scheduled trial assessments, the Investigator must determine the reasons and the circumstances as completely and accurately as possible.

In case a subject has to be withdrawn from the trial, the sponsor will be informed immediately. If there is a medical reason for withdrawal, the subject will remain under the supervision of the Investigator until satisfactory health has returned or the subject's health has reached a stable condition.

Subjects who are withdrawn from the trial after dosing will not be replaced.

In case of premature withdrawal from the trial, the processes outlined in Section 8.4.2 should be followed. In any case, the appropriate electronic Case Report Form (eCRF) section including the reason for discontinuation as defined in Section 8.6.2 must be completed.

The trial **can be** prematurely discontinued as described in Section 8.7.

### **6 TRIAL PARAMETERS**

### 6.1 Efficacy Endpoints

### 6.1.1 Primary Efficacy Endpoints

Two primary endpoints will be tested in the following order using hierarchical fixed sequence testing:

- 1. CFB in tCFS (NEI scale) at Day 29
- 2. CFB in Dryness Score (VAS) at Day 29

### 6.1.2 Key Secondary Efficacy Endpoints

The following key secondary efficacy endpoints will be evaluated:

- CFB in total conjunctival lissamine green staining score (Oxford scale) at Day 29
- Proportion of responders in cCFS score (≥ 1 score improvement on NEI scale) at Day 29
- Proportion of responders in tCFS score (≥ 3 scores improvement on NEI scale) at Day 29
- CFB in cCFS score (NEI scale) at Day 29
- CFB in tCFS score (NEI scale) at Day 15
- CFB in blurred vision (VAS) at Day 29






### **6.2** Safety Endpoints

- Visual acuity and CFB at each measured post-baseline visits;
- Slit-lamp biomicroscopy findings and CFB at each measured post-baseline visits;
- Intraocular pressure and CFB at each measured post-baseline visits;
- Dilated fundoscopy findings and CFB at each measured post-baseline visits;
- Systemic and ocular AEs




### 7 TRIAL MATERIALS

### 7.1 Investigational Medicinal Product(s)

### 7.1.1 <u>IMP(s)/ Formulation(s)</u>

### Run-In

• Systane Balance Lubricant Eye Drops

### Randomized IMPs

 Table 1.
 Active Investigational Medicinal Product

| Table 1. Metive investigational intenental frouter | |
|---|---|
| | Investigational Product |
| Product name: | CyclASol |
| Chemical name: | Cyclosporine A 0.1% |
| Dosage form: | |
| Unit dose: | |
| Route of administration: | Topical ocular administration |
| Physical description: | Colorless and clear ophthalmic solution |
| <b>Excipients:</b> | |
| Manufacturer: | |

 Table 2.
 Control/Reference Investigational Medicinal Product

| | Control/Reference Investigational Product |
|--------------------------|-------------------------------------------|
| Product name: | Vehicle (F4H5) |
| Chemical name: | |
| Dosage form: | |
| Unit dose: | |
| Route of administration: | Topical ocular administration |
| Physical description: | Colorless and clear ophthalmic solution |
| Excipients: | |
| Manufacturer: | |

### 7.1.2 <u>Labeling and Packaging of IMP</u>

For the run-in period, 1 bottle of Systane Balance will be labelled according to legal requirements.


As per the Code of Federal Regulations 21 part 312, section 312.6, the labels for the IMP shall be comprised of:

- Protocol number
- Investigational new drug statement
- Lot number
- Storage conditions
- Name and address of the sponsor

### 7.1.3 <u>IMP Storage</u>



### 7.1.4 Administration of run-in medication

At the end of Visit 0, qualified subjects will receive the run-in medication (Systane Balance). Their first dose of run-in medication will be in-office. They will then be instructed to dose at home BID up to and including the morning of Visit 1

Subjects will be instructed to dose in the morning and in the evening at bedtime. Subjects will record in the subject's diary that their doses were taken. At Visit 1, used/unused run-in will be collected from subjects.

### 7.1.5 <u>IMP Dispensation</u>




In case the subject needs a replacement bottle of IMP, the next bottle from the kit will be dispensed. If no bottle remains in the kit, a new kit will be assigned to the subject using IRT.

At Visit 3 remaining IMP will be collected from subjects for drug accountability.

### 7.1.6 Instructions for Use and Administration

Subjects will be instructed to instill one drop in each lower eyelid two times daily (in the morning and in the evening before bed). Subjects will be instructed to use a second drop only if the first drop misses the eye. Subjects will receive detailed written instructions how to store and dose IMP, and how to complete their diary.

Subjects will be instructed to immediately contact the site if there is any problem with the IMP or run-in medication (e.g. if the bottle was dropped or lost).

### 7.2 IMP Accountability

The investigator must keep an accurate accounting of IMP received from the supplier by maintaining a detailed inventory. This includes the amount of IMP received by the site, amount dispensed to subjects, amount of IMP returned to the investigator by the subjects, and the amount returned to the sponsor or designee upon the completion of the trial.

Investigational trial medication orders, records of receipts, dispensing records, and inventory forms will be examined and reconciled by designated site personnel. At each visit, subjects will return all bottles to designated site personnel for accountability purposes. Accountability will be ascertained by performing reconciliation between the amount of IMP cartons (kits and their components) sent to the site, the amount used and unused at the time of reconciliation. No investigative drugs or kits will be discarded prior to full accountability by sponsor's monitor.

### 7.3 IMP Handling and Disposal

Unless otherwise directed, at the end of the trial all returned used and unused IMP must be shipped from the clinical site to the depot for disposal of medications.

Note: The medications should not be disposed prior to full accountability by the sponsor's designated monitor.

The clinical site will provide a copy of all completed drug disposition forms to the sponsor after the completion of the trial.

### 7.4 Other Trial Supplies

Diaries, questionnaires, VAS rulers, Schirmer's test strips, sodium fluorescein, lissamine strips, Fluress, Tropicamide, Urine pregnancy tests.


### 8 TRIAL METHODS AND PROCEDURES

### 8.1 Concurrent Medications and Therapies

Therapy considered necessary for the subject's welfare that will not interfere with the evaluation of the study medication may be given at the discretion of the Investigator. If there is any question as to whether the medication may interfere, the Investigator should contact the Medical Monitor or Sponsor. Whenever possible, medications should be administered in dosages that remain constant throughout the study duration.

The use of any concurrent medication, prescription or over-the-counter, is to be recorded on the subject's source document and corresponding eCRF along with the reason the medication was taken.

### 8.2 Prohibited Medications

### 8.3 Restrictions and Prohibitions




### 8.4 Examination Procedures

### 8.4.1 <u>Procedures to be performed at Each Trial Visit with Regard to Trial Objective(s)</u>

The procedures outlined in this section will performed as described in Appendix 2: Examination Procedures, Tests, Equipment, and Techniques.

### Visit 0 (Day -14 $\pm$ 2 days): Screening

- Informed consent / HIPAA
- Medical/medication history and demographic data
- Review of qualification criteria (in-/exclusion criteria)
- Urine pregnancy test for females of childbearing potential
- Dryness Score (VAS)
- •
- Visual acuity (ETDRS)
- Slit-lamp biomicroscopy
- Fluorescein staining (NEI scale)
- Lissamine green staining (Oxford scale)
- Intraocular pressure
- Dilated fundoscopy
- In-office instillation of run-in drops to qualified subjects
- Dispensation of subject diary and run-in
- Non-leading AE questioning
- Qualified subjects are scheduled for Visit 1

### Visit 1 (Day 1): Baseline / Randomization

• At the beginning of the visit the subject will be asked about the time of last dose.

- Medical/Medication history update/Non-leading AE questioning
- Review of qualification criteria
- Dryness Score (VAS)




### Visit 2 (Day 15 $\pm$ 2): 2-Week Follow-Up

At the beginning of the visit the subject will be asked about the time of last dose.



- Visual acuity (ETDRS)
- Slit-lamp biomicroscopy
- Fluorescein staining (NEI scale)
- Lissamine green staining (Oxford scale)
- In-office instillation of randomized IMP (2<sup>nd</sup> dose of the day)
- Non-leading AE questioning
- Schedule for Visit 3


### Visit 3 (Day 29 $\pm$ 2): 4-Week Follow-Up and Trial Exit or ET

- At the beginning of the visit the subject will be asked about the time of last dose.
- Collection and review of IMP and subject diary;
- Medical/Medication history update/Non-leading AE questioning
- Urine pregnancy test for females of childbearing potential
- Dryness Score (VAS)
- •
- Visual acuity (ETDRS)
- Slit-lamp biomicroscopy
- Fluorescein staining (NEI scale)
- Lissamine green staining (Oxford scale)
- Elisamine green staming (Oxford Searc)
- Intraocular pressure
- Dilated fundoscopy
- Non-leading AE questioning
- Trial exit

### 8.4.2 Early Termination/Discontinuations

The following data from subjects discontinuing before randomization will be captured in the eCRF:

- Demographics
- AEs / SAEs
- Reason for discontinuation

Randomized and dosed subjects who discontinue treatment for any reason will be encouraged to undergo all subsequent trial visits and assessments.

Data from subjects discontinuing after randomization will be captured completely in the eCRF including Early Termination Visit and reason for discontinuation.

If a randomized subject is discontinued from the trial before Visit 3 (Day  $29 \pm 2$  days) and is not willing to perform all subsequent visits and assessments, all evaluations of Visit 3 (at least all


safety related evaluations) should be performed at Early Termination Visit on the day of early termination/discontinuation or at the discretion of the investigator.

### 8.4.3 Unscheduled Visits

An unscheduled visit may be performed during the course of the trial to ensure subject safety. All procedures performed at an unscheduled visit will be recorded in the source documents and on the Unscheduled Visit eCRF pages. Any unscheduled visit procedure listed in the eCRF that is not performed should be indicated as "not done."

Evaluations that may be conducted at an Unscheduled Visit include:

- Slit-lamp biomicroscopy;
- Visual acuity;
- Intraocular pressure;
- Urine pregnancy test (for women of childbearing potential);
- Dilated fundoscopy;
- Assessment of AEs:
- Assessment of concomitant medications and/or treatments; and
- Any other assessments needed in the judgement of the investigator.

### 8.5 Compliance with Dosing/Protocol Deviations

Subjects will be instructed on the proper use and storage of the IMP at Visits 0, 1 and 2 and provided with written instructions. Subject diaries and IMP will be collected at each visit from Visit 1 up to and including Visit 3 to assess subject compliance with the protocol.

A protocol deviation is any noncompliance with the clinical study protocol, GCP, or Study Operations manual requirements. The noncompliance may be on the part of the subject, the PI, or study staff. The Investigator should not deviate from the requirements of this protocol without prior written approval of the Medical Monitor or Sponsor/CRO, with the exception of a medical emergency. As a result of deviations, corrective actions may need to be developed by the study staff and implemented promptly.

All deviations from the protocol must be addressed in study subject source documents and promptly reported to the IRB according to their requirements. Protocol deviations will be assessed before DB lock as major or minor.

In case of a positive SARS-CoV-2 (COVID-19) test result or infection the subject must not undergo visits in the clinic until he/she is considered not to be infectious anymore. Potential skipped or delayed visits must be recorded as protocol deviations and denoted to be COVID-19


related. For those subjects, a Trial Exit Visit - also at a later point - is recommended if their health state allows.

### 8.6 Subject Disposition

### 8.6.1 Completed Subjects

A completed subject is one who has not been discontinued from the trial.

### 8.6.2 Discontinued Subjects

Notification of a subject's discontinuation and the reason for discontinuation will be made to and/or Novaliq and will be clearly documented on the eCRF as:

- Adverse Events;
- Protocol violations;
- Lack of efficacy;
- Administrative reasons (e.g., inability to continue, lost to follow up);
- Sponsor termination of trial;
- Subject choice (e.g. withdrawal of consent)
- Other

Discontinuations that are the direct result of SARS-CoV-2 (COVID-19) will be classified separately and clearly documented in the eCRF. A separate field will be completed to denote a COVID-19 related discontinuation and the specific reason will be documented utilizing the above noted list of subcategories.

Subjects must be discontinued as outlined in Section 5.5.

Subjects, who discontinue for any reason after randomization will not be replaced.

### 8.7 Trial Termination

The whole trial may be discontinued prematurely in the event of any of the following:

- New information leading to unfavorable risk-benefit judgment of the IMP, e.g. due to:
  - Occurrence of significant previously unknown adverse reactions or unexpectedly high intensity or incidence of known adverse reactions
  - Other unfavorable safety findings.
- Sponsor's decision that continuation of the trial is unjustifiable for medical or ethical reasons.
- Poor enrollment of subjects making completion of the trial within an acceptable time frame unlikely.
- Discontinuation of development of the sponsor's IMP.
- Terminated or suspended upon request of Health Authorities.


Novaliq GmbH Version 4.0. 15<sup>th</sup> March 2021

Health Authorities and Institutional Review Boards (IRBs)/ Independent Ethics Committees (IECs) will be informed about the discontinuation of the trial in accordance with applicable regulations.

### 8.8 Trial Duration

An individual subject's participation will involve four visits over approximately a 6-week period. After the trial, subjects will be treated according to the standard of care at the discretion of the treating physician. The total duration of the trial from "first subject in" to "last subject out" is expected to be 8 months.

Subjects who completed trial CYS-004 without major protocol deviations, have been compliant with CYS-004 trial procedures and application of IMP may be invited to enroll into an extension trial, CYS-005. CYS-005 will be a 12-months open-label safety extension trial of CYS-004 to assess the safety of topical CyclASol 0.1% for the treatment of DED.


#### 9 ADVERSE EVENTS

#### 9.1 Adverse Event

An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not the event is considered drug-related. An AE can therefore be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease occurring after the subject signed informed consent.

If there is a worsening of a medical condition that was present prior to the administration of the IMP or the run-in medication, this should also be considered a new AE and reported. Any medical condition present prior to the administration of the IMP or the run-in medication that remains unchanged or improved should not be recorded as an AE at subsequent visits.

Worsening of DED will be considered an AE only if the dry eye status of the subject exceeds their previous experiences with the condition. This will be determined by the subject and the investigator.

A clinically relevant worsening of visual acuity from screening visit (Visit 0). will be considered an AE.

IMP includes the investigational drug under evaluation and any comparator drug, vehicle, or any other medications required by the protocol given during any stage of the trial.

Documentation regarding the AE should be made as to the nature, date of onset, end date, severity, relationship to IMP, expectedness, action(s) taken, seriousness, and outcome of any sign or symptom observed by the physician or reported by the subject upon non-leading questioning.

AEs (both elicited and observed) will be monitored from the time of signing informed consent throughout the trial. All AEs will be promptly reviewed by the investigator for accuracy and completeness. All AEs will be documented on the appropriate source document and eCRF.

#### 9.1.1 Severity

Severity of an AE is defined as a qualitative assessment of the degree of intensity of an AE as determined by the investigator or reported to him/her by the subject. The assessment of severity is made irrespective of relationship to investigational product or seriousness of the event and should be evaluated according to the following scale:

- *Mild*: Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- *Moderate*: Event is bothersome, possibly requiring additional therapy, and may interfere with the subject's daily activities.
- Severe: Event is intolerable, necessitates additional therapy or alteration of therapy, and interferes with the subject's daily activities.


Severity is not the same as "seriousness", which is based on the outcome or action criteria usually associated with events that pose a threat to life or functioning (see Section 9.2). Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

## 9.1.2 Relationship to Investigational Product

The relationship of each AE to the IMP should be determined by the investigator using these explanations:

- *Suspected*: A reasonable possibility exists that the investigational product caused the AE.
- *Not Suspected*: A reasonable possibility does not exist that the investigational product caused the AE.

Suspected adverse reaction means any AE for which there is a reasonable possibility that the investigational product caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the IMP and the AE. Types of evidence that would suggest a causal relationship between the IMP and the AE include: a single occurrence of an event that is uncommon and known to be strongly associated with IMP exposure (e.g., angioedema, hepatic injury, Stevens-Johnson Syndrome); one or more occurrences of an event that is not commonly associated with IMP exposure, but is otherwise uncommon in the population exposed to the IMP (e.g., tendon rupture); an aggregate analysis of specific events observed in a clinical trial (such as known consequences of the underlying disease or condition under investigation or other events that commonly occur in the trial population independent of drug therapy) that indicates those events occur more frequently in the IMP-treatment group than in a concurrent or historical control group.

#### 9.1.3 <u>Expectedness</u>

The expectedness of an AE should be determined based upon existing safety information about the IMP. CyclASol contains the active ingredient CsA and the vehicle F4H5 and has been tested in three clinical studies up to now, and AEs of those have been listed in the Investigator's Brochure. Therefore, the following definition will be used:

- *Unexpected*: An AE that is not listed in the investigator's brochure (IB) in the Adverse Reaction Section at the specificity or severity that has been observed.
- Expected: An AE that is listed in the investigator's brochure (IB) in the Adverse Reaction Section at the specificity and severity that has been observed.
- *Not Applicable*: Any AE that is unrelated to the IMP.

The Investigator should initially classify the expectedness of an AE, but the final classification is subject to the sponsor's determination.

#### 9.1.4 Outcome

The outcome of any AE will be determined and recorded using the following categories:


- Recovered/Resolved
- Recovering/Resolving
- Not Recovered/Not Resolved
- Recovered/Resolved with Sequelae
- Lost to Follow-up
- Fatal
- Unknown

#### 9.1.5 <u>Period of Observation</u>

For the purpose of this study, the period of observation for collection of adverse events extends from the time the patient gives informed consent until the end of the Visit 3 at (Day  $29 \pm 2$ ) or Early Termination.

If the investigator detects a Serious Adverse Event (see Section 9.2) in a study patient after the end of the period of observation this should be reported to the Sponsor only if the investigator considers the event related to prior study treatment or procedures. The investigator should contact the sponsor to determine how the adverse event should be documented and reported.

#### 9.2 Serious Adverse Events

An AE is considered serious if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death;
- A life-threatening AE;
  - O Note: An AE is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the subject or subject at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death.
- Inpatient hospitalization or prolongation of existing hospitalization;
  - O Note: The term "inpatient hospitalization" refers to any inpatient admission (even if less than 24 hours). For chronic or long-term inpatients, inpatient admission includes transfer within the hospital to an acute/intensive care inpatient unit. Inpatient hospitalization does not include: emergency room visits; outpatient/same-day/ambulatory procedures; observation/short stay units; rehabilitation facilities; hospice facilities; nursing homes; or clinical research/phase 1 units.
  - O Note: The term "prolongation of existing hospitalization" refers to any extension of an inpatient hospitalization beyond the stay anticipated or required for the reason for the initial admission as determined by the investigator or treating physician.
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;


- O Note: A serious adverse event (SAE) specifically related to visual threat would be interpreted as any potential impairment or damage to the subject's eyes (e.g., hemorrhage, retinal detachment, central corneal ulcer or damage to the optic nerve).
- A congenital anomaly/birth defect;
- Medically important.
  - Note: Important medical events that may not result in death, are life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

| 9. | 3 | <b>Procedures</b> | for | Reporting | Adverse | <b>Events</b> |
|----|---|-------------------|-----|-----------|---------|---------------|
| - | _ | | | | | |

| All AEs and their outcomes must be reported to Novaliq, |
|---|
| and the IRB as required by the IRB, federal, state, or local regulations and governing |
| health authorities and recorded on the appropriate eCRF. |
| 9.3.1 Reporting a Serious Adverse Event |
| To ensure subject safety, all SAEs, regardless of their relationship to the IMP, must be immediately reported (i.e. within a maximum 24 HOURS after becoming aware of the event). All information relevant to the SAE must be recorded on the appropriate SAE report forms. The investigator is obligated to pursue and obtain information requested by and/or Novaliq in addition to that information reported on the case report form. All subjects experiencing a SAE must be followed up and the outcome reported. |
| In the event of a SAE, the investigator must notify immediately; obtain and maintain in his/her files all pertinent medical records, information, and medical judgments from colleagues who assisted in the treatment and follow-up of the subject; provide and the trial sponsor with a complete case history, which includes a statement as to whether the event was or was not suspected to be related to the use of the IMP; and inform the IRB of the AE within their guidelines for reporting SAEs |

External safety service provider

Email:
Fax:

Contact information for Medical Monitor:

Medical Monitor:
Office Telephone:


Alternative Telephone (24-hr line):
Fax:

## 9.3.2 Reporting a Suspected Unexpected Serious Adverse Reaction

All SAE that are 'suspected reactions' and 'unexpected' are to be reported to the IRB/IEC as required by the IRB/IEC, federal, state, or local regulations and governing health authorities.

# 9.4 Procedures for Unmasking of IMP

All subjects, investigators, and trial personnel involved with the conduct of the trial will be masked with regard to treatment assignments. When medically necessary, the investigator may need to determine what treatment arm has been assigned to a subject.

In a medical emergency, when the management of a subject's condition requires knowledge of the treatment assignment, the Investigator, or designee, will obtain the trial treatment assignment from the IRT. If possible, the medical emergency should be discussed with the medical monitor prior to obtaining the treatment assignment, or as soon after as possible. The sponsor's external safety provider may unmask for regulatory submission determination of an SAE when necessary (see Section 9.3.1).

In a non-emergency situation, when a code break is required, it must be discussed with the medical monitor and/or and Novaliq. The code break must be approved in writing by the sponsor.

If the randomization code for a subject is broken, the Investigator will record the date and reason for lifting the mask for that subject in the source documents. Upon unmasking, the subject will be withdrawn from the trial and should complete both the Early Termination and Follow-up procedures.

## 9.5 Type and Duration of the Follow-up of Subjects after Adverse Events

The investigator will follow unresolved AEs to resolution until the subject is lost to follow-up or until the AE is otherwise classified. Resolution means the subject has returned to baseline state of health or the investigator does not expect any further improvement or worsening of the AE. If the subject is lost to follow-up, the investigator should make 3 reasonable attempts to contact the subject via telephone, post, or certified mail. All follow-up will be documented in the subject's source document. Non-serious AEs identified on the last scheduled contact must be recorded on the AE eCRF page with the status noted.

If the investigator becomes aware of any new information regarding an existing SAE (i.e., resolution, change in condition, or new treatment), a new SAE Report Form must be completed and e-mailed/ faxed to within 24 hours of the site's awareness of the new information. The original SAE form is not to be altered. The report should describe whether the event has resolved or continues and how the event was treated.


# 9.6 Procedures for Reporting Pregnancies

Pregnancy in itself is not considered an AE or SAE (unless there is a suspicion that an IMP may have interfered with the effectiveness of a contraceptive medication), but it is an important medical event that must be followed up. Any pregnancy that occurs during the clinical trial where the fetus could have been exposed to IMP must be followed through the outcome of the pregnancy.

It is the responsibility of the Investigator to obtain the outcome and condition of the infant information within 30 calendar days after the initial notification and approximately 30 calendar days postpartum.

If a subject or Investigator suspects that the subject may be pregnant prior to IMP administration, the IMP must be withheld until the results of pregnancy testing are available. If pregnancy is confirmed, the subject must not receive IMP and must not be enrolled in the study. If pregnancy is suspected while the subject is receiving IMP treatment, the IMP must immediately be withheld until the result of pregnancy testing is known.

If a female has a positive pregnancy test during the trial, then the investigator must report the pregnancy and the outcome of the pregnancy to within 24 hours of learning about the pregnancy.

A Pregnancy Reporting Form will be completed by the trial site's principal investigator and sent to via the SAE Fax number (see Section 9.3). will forward the documentation to the medical monitor, project manager and the sponsor for review.

At the completion of the pregnancy, the Pregnancy Outcome Form is to be submitted to the SAE contact details. Will manage the query and reconciliation process until the pregnancy documentation is complete.


## 10 STATISTICAL HYPOTHESES AND METHODS OF ANALYSES

## 10.1 Analysis Populations

The following analysis population will be considered:

- <u>Full Analysis Set (FAS)</u> The FAS includes all randomized subjects who received at least one dose of investigation product. The primary analysis will be performed on the FAS. Subjects in the FAS will be analyzed as randomized.
- Per Protocol Set (PPS) The PPS includes subjects in the FAS who do not have major protocol deviations and who complete the trial. Protocol deviations will be assessed prior to database lock and unmasking. The PPS will be analyzed using observed data only for efficacy variables. Subjects in the PPS will be analyzed as treated.
- <u>Safety Set (SAF)</u>—The SAF includes all randomized subjects who have received at least one dose of the investigational product. The SAF will be analyzed for all safety assessments. Subjects in the SAF will be analyzed as treated.

The statistical analysis of safety data will be performed for the SAF. The analysis of baseline and efficacy data will be performed for the FAS. The primary efficacy analyses will also be performed on the PPS as sensitivity analyses.

# 10.2 Statistical Hypotheses

The primary endpoints will be tested in a hierarchical fixed sequence in the following order. The statistical hypotheses for the primary endpoint of CFB in tCFS score (NEI scale) at Day 29 are as follows:

- $H_{01}$ : The difference, between study eyes treated with CyclASol and study eyes treated with vehicle, in the mean CFB in tCFS score (NEI scale) at Day 29 = 0.
- H<sub>A1</sub>: The difference, between study eyes treated with CyclASol and study eyes treated with vehicle, in the mean CFB in tCFS score (NEI scale) at Day  $29 \neq 0$ , with superiority claimed if the difference is less than 0 (CyclASol minus vehicle).

The statistical hypotheses for the primary endpoint of the CFB in Dryness Score (VAS) at Day 29 are as follows:

- $H_{02}$ : The difference, between subjects treated with CyclASol and subjects treated with vehicle, in the mean CFB in Dryness Score (VAS) at Day 29 = 0.
- $H_{A2}$ : The difference, between subjects treated with CyclASol and subjects treated with vehicle, in the mean CFB in Dryness Score (VAS) at Day  $29 \neq 0$ , with superiority claimed if the difference is less than 0 (CyclASol minus vehicle)

Hierarchical fixed sequence testing will be employed to maintain the type I error rate. The primary analyses will first test the difference in the mean CFB in tCFS score (NEI scale) between


treatments at Day 29. If the test of the difference is statistically significant at the two-sided alpha = 0.05 level in favor of CyclASol, then the trial will be considered a success; CyclASol will be declared to be superior to vehicle in the mean CFB in tCFS score (NEI scale) at Day 29; and the difference in the mean CFB in Dryness Score (VAS) between treatments at Day 29 will be tested at the two-sided alpha = 0.05 level.

If in addition to a statistically significant test of the difference in the mean CFB in tCFS score (NEI scale) at Day 29 in favor of CyclASol, the test of the difference in the mean CFB in Dryness Score (VAS) at Day 29 is also statistically significant in favor of CyclASol, then CyclASol will be declared to be superior to vehicle in both the mean CFB in tCFS score (NEI scale) and the mean CFB in Dryness Score (VAS) at Day 29.

# 10.3 Sample Size

The trial has been designed to have 90% power to reject both H<sub>01</sub> and H<sub>02</sub> assuming independence between the sign and symptom endpoint; positive correlation between these two endpoints would increase the overall power.

Three hundred seventy nine (379) full analysis set (FAS) subjects (study eyes) per treatment group yield 96.8% power to reject  $H_{01}$  in favor of  $H_{A1}$  and conclude superiority of CyclASol over vehicle in the mean CFB in tCFS score at Day 29 assuming a true difference (CyclASol minus vehicle) of -0.75, a common standard deviation of 2.7, and a two-sided alpha = 0.05.

Additionally, 379 FAS subjects per treatment group yield 93.0% power to reject  $H_{02}$  in favor of  $H_{A2}$  and conclude superiority of CyclASol over vehicle in the mean CFB in Dryness Score (VAS) at Day 29, assuming a true difference (CyclASol minus vehicle) of -5.0, a common standard deviation of 20.0, and a two-sided alpha = 0.05.

Therefore, assuming independence between tCFS score and Dryness Score (VAS), 379 FAS subjects per treatment group yields 96.8% \* 93.0% = 90.0% power to reject both H<sub>01</sub> and H<sub>02</sub>.

Accounting for subject discontinuations, approximately 834 total subjects (417 per treatment arm) will be enrolled

#### **10.4 Statistical Analysis**

#### 10.4.1 General Considerations

Quantitative variables will be summarized using number of subjects (n), mean, median, standard deviation, minimum and maximum. The dichotomous variables will be summarized using counts and percentages.

All summaries will be presented by treatment group. Summaries will be provided for demographics, baseline medical history, concurrent therapies, and subject disposition.


For the purpose of summarization, medical history, concurrent therapies, and AEs will be coded to MedDRA and WHO Drug dictionaries, as appropriate.

Baseline measures are defined as the last non-missing measure prior to the initiation of randomized study treatment. CFB will be calculated as Visit – Baseline.

For observed measures obtained on Visit 3 more than + 7 days out of window for any reason, measures will be considered missing data for all efficacy analyses and not used for analyses unless otherwise specified.

## 10.4.2 Unit of Analysis

For efficacy endpoints, the unit of analysis will be the "study eye" as defined by the following:

| • | · |
|---|---|

# 10.4.3 Missing Data

| The primary analysis will be completed with available data per subject from the Full Analysis Set (FAS) using Estimand 1, assuming the rate of missing data for an endpoint is <5%. |
|---|




### 10.4.4 Multiplicity Considerations

Hierarchical sequence testing will be employed to maintain the type I error rate. The primary analyses will first test the difference in the mean CFB in tCFS score (NEI scale) between treatments at Day 29. If the test of the difference is statistically significant at the two-sided alpha = 0.05 level in favor of CyclASol, then the trial will be considered a success; CyclASol will be declared to be superior to vehicle in the mean CFB in tCFS score (NEI scale) at Day 29; and the difference in the mean CFB in Dryness Score (VAS) between treatments at Day 29 will be tested at the two-sided alpha = 0.05 level.

If in addition to a statistically significant test of the difference in the mean CFB in tCFS score (NEI scale) at Day 29 in favor of CyclASol, the test of the difference in the mean CFB in Dryness Score (VAS) at Day 29 is also statistically significant in favor of CyclASol, then CyclASol will be declared to be superior to vehicle in both the mean CFB in tCFS score (NEI scale) and the mean CFB in Dryness Score (VAS) at Day 29.

Additionally, the key secondary efficacy endpoints will be alpha adjusted using the following composite methodology:

The following key secondary endpoints will be tested hierarchically:

- 1. CFB in total conjunctival lissamine green staining score (Oxford scale) at Day 29
- 2. Proportion of responders in cCFS score ( $\geq 1$  score improvement on NEI scale) at Day 29)
- 3. Proportion of responders in tCFS ( $\geq$  3 score improvement on NEI scale) at Day 29
- 4. CFB in cCFS score (NEI scale) to Day 29


Inference will only be made on these endpoints, at a 2-sided alpha = 0.05, if both primary endpoints and any higher order key secondary endpoints are statistically significant at a 2-sided alpha = 0.05 in favor of CyclASol.

If all four of these key secondary endpoints and both primary endpoints demonstrate statistical significance at a 2-sided apha = 0.05 in favor of CyclASol, then the following two key secondary endpoints will be tested simultanteously using Hochberg's procedure to maintain an overall two-sided alpha = 0.05:

- CFB in visual analogue scale (VAS) for blurred vision and at Day 29
- CFB in tCFS (NEI scale) at Day 15

Hochberg's procedure will be implemented by ordering the two-sided p-values from these three key secondary endpoints from highest to lowest. Each of these ordered p-values will be tested against 0.05 \* [(3 - k)/2] where 2 is the number of key secondary endpoints tested, 3 is the number of key secondary endpoints + 1, and k is the rank order of the endpoint. If the first ordered endpoint (highest to lowest) has a two-sided p-value < 0.05 in favor of CyclASol then both endpoints will be considered statistically significant. If the first ordered endpoint does not have a two-sided p-value < 0.05 in favor of CyclASol, then the two-sided p-value for the second ordered endpoint will be compared against 0.025.

## 10.4.5 Primary Efficacy Analyses

The primary comparisons in this trial will be between CyclASol versus vehicle at Day 29 in the FAS with available data per subject using the following estimand:




Analyses based on Estimand 2 and Estimand 3 will be additional sensitivity analyses.






The primary efficacy endpoints (e.g. CFB in tCFS score [NEI scale] and Dryness Score [VAS]) will be analyzed separately using an ANCOVA model with terms for baseline value and treatment.

Least squares mean for each treatment group and for the difference between treatment groups will be presented from the model together with two-sided p-values and 95% confidence intervals.

| Two-sample t-tests and Wilcoxon rank sum tests comparing treatment groups will be performed |
|---|


#### 10.4.6 Key Secondary Efficacy Analyses

The following key secondary endpoints will be tested hierarchically:

- 1. CFB in total conjunctival lissamine green staining score (Oxford scale) at Day 29
- 2. Proportion of responders in cCFS score (≥ 1 score improvement on NEI scale) at Day 29)
- 3. Proportion of responders in tCFS score (≥ 3 score improvement on NEI scale) at Day 29
- 4. CFB in cCFS score (NEI scale) to Day 29

Inference will only be made on these endpoints, at a 2-sided alpha = 0.05, if both primary endpoints and any higher order key secondary endpoints are statistically significant at a 2-sided alpha = 0.05 in favor of CyclASol.

If all four of these key secondary endpoints and both primary endpoints demonstrate statistical significance at a 2-sided apha = 0.05 in favor of CyclASol, then the following two key secondary endpoints will be tested simultanteously using Hochberg's procedure (Section 10.4.4) to maintain an overall two-sided alpha = 0.05:

- CFB in VAS for blurred vision and at Day 29
- CFB in tCFS (NEI scale) at Day 15

Quantitative key secondary efficacy endpoints will be summarized similarly to the primary effiacy endpoints.

Dichotomous key secondary endpoints (proportion of responders) will be summarized descriptively (frequency and percentage) and analyzed using a logistic regression model with terms for baseline value and treatment. Least squares mean for each treatment group and for the difference between treatment groups will be presented from the model together with two-sided p-values and 95% confidence intervals. Pearson chi-squared analysis comparing the treatment groups will be performed as sensitivity analyses.






# 10.4.9 <u>Safety Variables Analyses</u>

All safety analyses will be performed on the Safety Population.

Dosing information for each treatment and each subject will be listed. Discontinuation of treatment will be summarized by treatment received. The primary reason for trial drug discontinuation will also be summarized by treatment received.


Adverse events (AEs) will be coded using the MedDRA dictionary. Frequencies and percentages of treatment-emergent adverse events (TEAEs) will be summarized at the subject level by system organ class and preferred term for all TEAEs, treatment related TEAEs, serious TEAEs, and TEAEs causing premature discontinuation by treatment group. An AE is treatment emergent if it occurs or worsens after the first dose of trial treatment. Similar summaries will be presented for all TEAEs by maximal severity. Separate summaries will be performed for ocular and non-ocular AEs.

Concomitant medications will be coded using the most recent version of WHO-Drug Dictionary and summarized by treatment group.

Other safety endpoints including visual acuity, slit lamp biomicroscopy, intraocular pressure (IOP) and dilated fundoscopy will be summarized by treatment group and visit using descriptive statistics. Changes or shifts from baseline will also be summarized where appropriate. For assessments performed by eye, study eye and fellow eye will be summarized separately. In addition, changes from baseline to worst on-treatment value for ocular safety assessments will be summarized.

#### 10.4.10 Interim Analyses

No interim analyses are planned for this trial.

# 10.5 Additional Analyses






# 11 COMPLIANCE WITH GOOD CLINICAL PRACTICES, ETHICAL CONSIDERATIONS, AND ADMINISTRATIVE ISSUES

This trial will be conducted in compliance with the protocol, current Good Clinical Practices (GCPs), including the International Conference on Harmonization (ICH) Guidelines, and in general, consistent with the Declaration of Helsinki. In addition, all applicable local, state, and federal requirements relevant to the use of investigational products in the countries involved will be adhered to.

# 11.1 Protection of Human Subjects

## 11.1.1 Subject Informed Consent

Informed consent/assent must take place before any trial specific procedures are initiated. Signed and dated written informed consent must be obtained from each subject prior to performing any trial specific procedures and assessments.

All informed consent/assent forms must be approved for use by the sponsor and receive approval/favorable opinion from an IRB prior to their use. If the consent form requires revision (e.g., due to a protocol amendment or significant new safety information), it is the investigator's responsibility to ensure that the amended informed consent is reviewed and approved by the governing IRB and that it is read, signed and dated by all subjects subsequently enrolled in the trial as well as those currently enrolled in the trial.

#### 11.1.2 Institutional Review Board (IRB) Approval

This trial is to be conducted in accordance with Institutional Review Board regulations (U.S. 21 CFR Part 56.103).

Only an IRB/IEC approved version of the informed consent form will be used.

## 11.2 Ethical Conduct of the Trial

This trial will be conducted in accordance with the ethical principles that originated with the Declaration of Helsinki.


# 11.3 Subject Confidentiality

All personal trial subject data collected and processed for the purposes of this trial should be maintained by the investigator and his/her staff with adequate precautions as to ensure that the confidentiality of the data in accordance with local, state, and federal laws and regulations.

Monitors, auditors and other authorized representatives of the sponsor, the IRB/IEC approving this trial, the FDA, the Department of Health and Human Services, other domestic government agencies, and other foreign regulatory agencies will be granted direct access to the trial subject's original medical and trial records for verification of the data and/or clinical trial procedures. Access to this information will be permitted to the aforementioned individuals to the extent permitted by law.

A report of the results of this trial may be published or sent to the appropriate health authorities in any country in which the investigational product may ultimately be marketed, but the subject's identity will not be disclosed in these documents.

#### 11.4 Documentation

Source documents may include a subject's medical records, hospital charts, clinic charts, the investigator's trial subject files, as well as the results of diagnostic tests such as X-rays, laboratory tests, and ECGs. The investigator's copy of the eCRFs serves as the investigator's record of a subject's trial-related data.

## 11.4.1 Retention of Documentation

All trial related correspondence, subject records, consent forms, record of the distribution and use of all investigational products and copies of case report forms should be maintained on file for at least two years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region; or until at least two years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the sponsor. It is the responsibility of the sponsor to inform the investigator/institution as to when these documents no longer need to be retained. The investigator must notify the sponsor prior to destroying trial documentation even after the above-mentioned time has passed.

If the responsible investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping trial records, custody must be transferred to a person who will accept the responsibility. The sponsor must be notified in writing of the name and address of the new custodian.


# 11.5 Recording of Data on Source Documents and Electronic Case Reports Forms (eCRFs)

All subject data will be captured in the subject source documents which will be transcribed to the eCRFs. The investigator is responsible for ensuring that trial data is completely and accurately recorded on each subject's eCRF, source document, and all trial-related materials. All trial data should also be attributable, legible, contemporaneous, and original. Recorded data should only be corrected in a manner that does not obliterate, destroy, or render illegible the previous entry (e.g., by drawing a single line through the incorrect entry and writing the revision next to the corrected data). An individual who has corrected a data entry should make clear who made the correction and when, by adding to the correction his/her initials as well as the date of the correction.

Data entry of all enrolled and randomized subjects will use software that conforms to 21 CFR Part 11 requirements and will be performed only by staff that have been trained on the system and have access to the system. For screen failure subjects, the following data will be entered: AE, SAE, demographics and reason for screen failure. An audit trail will be maintained within the electronic system to capture all changes made within the eCRF database. After the end of the trial and database lock, compact discs (CDs) containing copies of all applicable subjects' eCRFs will be provided to each investigator site to be maintained on file by the investigator.

# 11.6 Monitoring and Quality Assurance

During the course of the trial a clinical research associate (CRA) will make routine site visits to review protocol compliance, assess IMP accountability, and ensure the trial is being conducted according to the pertinent regulatory requirements. The review of the subjects' medical records will be performed in a manner that adequately maintains subject confidentiality. Further details of the trial monitoring will be outlined in a monitoring plan.

Domestic and foreign regulatory authorities, quality assurance, sponsor and or its designees may carry out on-site inspections and/or audits which may include source data checks. Therefore, direct access to the original source data will be required for inspections and/or audits. All inspections and audits will be carried out with consideration to data protection as well as subject confidentiality to the extent that local, state, and federal laws apply.

# 11.7 Handling of Biological Samples

Not applicable.

#### 11.8 Publications

Authorship and manuscript composition will reflect cooperation among all parties involved in the trial. Authorship will be established before writing the manuscript. The trial sponsor will have the final decision regarding authorship, manuscript and publication.


#### 12 REFERENCES

Agarwal P, Khun D, Krösser S, Eickhoff K, et al. Preclinical studies evaluating the effect of semifluorinated alkanes on ocular surface and tear fluid dynamics. *Ocular Surf.* 2019 Apr;17(2): 241-249

Benitez-del-Castillo J, Labetoulle M, Baudouin C, et al. Visual acuity and quality of life in DED: Proceedings of the OCEAN group meeting. *The Ocular Surface 2017; 15*: 169-178.

Craig JP, Nichols KK, Nichols JJ, Caffrey B, Dua HS, Akpek EK, Tsubota K, Joo CK, Liu Z, Nelson JD, Stapletin F. TFOS DEWS II definition and classification report. The Ocular Surface 2017: 276-283.

Krafft MP, Riess JG. Chemistry, physical chemistry, and uses of molecular fluorocarbon-hydrocarbon diblocks, triblocks, and related compounds - unique "apolar" components for self-assembled colloid and interface engineering. *Chem Rev* 2009; 109: 1714-92.

Le Q, Zhou X, Ge L, Wu L, Hong J, Xu J. Impact of dry eye syndrome on vision-related quality of life in a non-clinic-based general population. *BMC Ophthalmology* 2012; 12(22): 1-8

Lemp MA. Report of the National Eye Institute/Industry Workshop on Clinical Trials in Dry Eyes. *CLAO J.* 1995; 21(4): 221-232.

Lin PY, Tsai SY, Cheng CY, Liu JH, Chou P, Hsu WM. Prevalence of dry eye among an elderly Chinese population in Taiwan: the Shihpai Eye Trial. *Ophthalmology* 2003; 110(6):1096-101.

McCarty CA, Bansal AK, Livingston PM, Stanislavsky YL, Taylor HR. The epidemiology of dry eye in Melbourne, Australia. *Ophthalmology* 1998; 105(6):1114-9.

Novack GD, Penny A, Barabino S, Bergamini MVW, Ciolino JB, Foulks GN, Goldstein M, Lemp MA, Schrader S, Woods C, Stapleton F. TFOS DEWS II Clinical Trial Design Report. *The Ocular Surface* 2017: 635-655.

Pflugfelder SC, de Pavia CS. The pathophysiology of dry eye disease. What we know and future directions for research. *Ophthalmology* 2017; 124: S4-S13.

Schaumberg DA, Sullivan DA, Dana MR. Epidemiology of dry eye syndrome. *Adv Exp Med Biol* 2002; 506, 989-98.

Schaumberg DA, Dana R, Buring JE, Sullivan DA. Prevalence of dry eye disease among US men: estimates from the Physicians' Health Studies. *Arch Ophthalmol* 2009; 127: 763-8.

Schaumberg DA, Sullivan DA, Buring JE, Dana MR. Prevalence of dry eye syndrome among US women. *Am J Ophthalmol* 2003; 136: 318-26.


Schiffman RM, Walt JG, Jacobsen G, Doyle JJ, Lebovics G, Sumner W. Utility Assessment among patients with dry eye disease. *Ophthalmology* 2003; 110: 1412-1419

Van Setten G, Labetoulle M, Baudouin C, Rolando M. Evidence of seasonality and effects of psychometry in dry eye disease. *Acta Ophthalmol*. 2016: 1-8.

